CLINICAL TRIAL: NCT03063385
Title: Testing a Latino Web-based Parent-adolescent Sexual Communication Intervention
Brief Title: Puerto Rico Cuidalos Parent-adolescent Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of Puerto Rico (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 820216; 7R01NR013505 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2017-02-24 (Actual); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: HIV/AIDS and Infections; Sexually Transmitted Diseases; Pregnancy Prevention
Keywords: Adolescents; Parents; Web-based; Puerto Rico; Latino; Sexual communication; Stigma; Randomized controlled trial; STD; Intercourse; Sexual behavior; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Sexually Transmitted Diseases; Social Stigma; Coitus; Sexual Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parental communication intervention (Experimental): The parental experimental intervention consists of a 60-minute web-based intervention consisting of several modules.
  Interventions: Behavioral: Parental Communication intervention
- Health promotion control condition. (Active Comparator): The Health promotion control condition will be web-based and provide useful information for Puerto Rican parents and youth.
  Interventions: Behavioral: Health promotion control condition

INTERVENTIONS:
Behavioral: Parental Communication intervention — In this intervention, we focus on providing parents with basic knowledge about pregnancy, HIV/AIDS, and STDs as a basis for effectively communicating with their adolescents. We work to support attitudes and develop skills to facilitate communication in general and specifically sexual communication. Based on our prior work we focus on prevention beliefs, reaction beliefs, and communication efficacy. Importantly, we include a component on HIV/AIDS stigma as we conceptualize this to impact attitudes and communication about sex. We will program the intervention in such a way so that parents will have to view the Cuídalos program sequentially and in its totality before being able to review any content.
  Arms: Parental communication intervention
Behavioral: Health promotion control condition — In this intervention, we provide a web-based program relying on existing Spanish language web-sites to provide participants with helpful information to prevent significant health problems affecting Puerto Rican adolescents that are related, not to sexual behavior, but to other behaviors. Similar to the experimental condition, we will develop a set of "homework" related to diet and exercise that we will ask parents to complete with their adolescents.
  Arms: Health promotion control condition.

SUMMARY:
Latino adolescents are at high risk for HIV/AIDS, other sexually transmitted infections (STIs), and unintended pregnancies. Puerto Rican adolescents, in particular, experience disparities in these areas, yet few adolescent and even fewer parent interventions have been developed to address these important issues with this underserved population. Parent-adolescent programs are an effective approach to reduce adolescent sexual risk behavior and associated negative consequences. A web-based parent communication intervention provides an opportunity to strengthen and enhance programs that are designed for adolescents by providing additional support for safer sex decisions, and to increase parents' access to sexual health education programs by decreasing barriers that keep them from participating in these interventions (e.g., low cost, can be viewed privately, at parents convenience, minimizes competing time with work and family). The purpose of this proposed study is to evaluate a brief theoretically informed (i.e., Ecodevelopmental Theory, Theory of Reasoned Action/Planned Behavior, Social Cognitive Theory 1-6), culturally appropriate, and linguistically tailored web-based parental communication program, Cuídalos ("Take care of them"), designed to improve parent-adolescent sexual communication and reduce adolescent sexual risk behavior. Recent findings from an NIH funded R21 randomized control trial (RCT) testing a brief computer-based version of the Cuídalos program indicated that the program increased parent-adolescent general communication and sexual risk communication with English and Spanish speaking U.S. Latinos. Further, despite limited or no previous computer use, parents reported they liked and learned from the program, and that it was easy to use and accessible.

DETAILED DESCRIPTION:
In this proposed RCT, and based on recommendations from parents who participated in the initial Cuídalos7 intervention trial, the investigators plan to modify the program by: 1) increasing the amount of content related to sexual communication (e.g., more case studies and interactive activities); 2) adding a module on stigma (towards HIV/AIDS); 3) increasing access by moving from a computer-based to a web-based platform; and 4) increasing the flexibility in how the program is used (e.g., ability to view the entire program or specific modules more than once). In order to examine the efficacy of the program, the investigators will recruit 680 parents and one of the participant's adolescents from schools, community-based and governmental organizations in Puerto Rico, and will randomly assign parents to receive: 1) the Cuídalos intervention; or 2) a web-based health promotion control intervention focused on the prevention of diabetes and cardiovascular disease. Parents and adolescents will complete measures at pre-intervention and at 3- (parents only), 6-, and 12 month follow-ups.

The investigators will address the five following specific aims:

1. Determine whether the Cuídalos intervention increases parents' comfort with, as well as the amount of, general and sexual risk-specific communication with adolescents and whether it decreases stigma (towards HIV/AIDS) at 3-,6-, and 12- month follow-ups as compared to the general health promotion control intervention.
2. Determine whether the Cuídalos intervention decreases self-reported adolescent intercourse and unprotected intercourse at 6-, and 12- month follow-ups as compared to the general health promotion control intervention.
3. Identify theory-based variables (e.g., attitudes, subjective norms, perceived behavioral control, and intentions) that mediate the intervention effects of Cuídalos on parents' self-reported comfort with and amount of communication with their adolescents.
4. Determine whether the effects of the Cuídalos intervention on adolescents sexual behavior and parent adolescent communication are moderated by individual (adolescents: sexual experience, gender, age, stigma; parents: gender, age, computer access and experience, frequency and time engaged in the program), and microsystem (adolescents: parent-adolescent communication) factors.
5. Examine the cost-effectiveness of the web-based Cuídalos intervention on adolescent sexual behavior.

Results from this study will inform the use and efficacy of a web-based Cuídalos program for Puerto Rican parents. This study is an innovative and timely effort given the existing disparities in sexual health outcomes among Latino youth, the lack of culturally and linguistically effective interventions for Latino parents and adolescents, and the absence of web-based interventions with Latinos. If the program is efficacious, the web-based format will accelerate the translation of this program into public health practice and will be an important contribution in supporting adolescent sexual health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* one parent and one son or daughter between 13 and 17 years of age must agree to be in the study
* in Puerto Rico

Exclusion Criteria:

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 660 (Actual)
Dates: Start 2012-09; Primary Completion 2016-08 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonia M Villarruel, PhD, RN, Principal Investigator — University of Pennsylvania; Nelson Varas-Diaz, PhD, Principal Investigator — University of Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villarruel AM, Loveland-Cherry CJ, Ronis DL. Testing the Efficacy of a Computer-Based Parent-Adolescent Sexual Communication Intervention for Latino Parents. Fam Relat. 2010 Dec 1;59(5):533-543. doi: 10.1111/j.1741-3729.2010.00621.x. PMID 21116466

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parental Communication Intervention | Health Promotion Control Condition.
Started | 330 | 330
3-month Follow-up | 257 | 259
6-month Follow-up | 265 | 259
12-month Follow-up | 243 | 254
Completed | 243 | 254
Not Completed | 87 | 76

BASELINE CHARACTERISTICS:
Population: A total of 660 parent/adolescent dyads (N=1,320) were randomized and met the following criteria: 1) agreed to engage in the study as a dyad, and 2) adolescent was between 13 and 17 years of age. We did not exclude parents or adolescents based on their literacy or computer literacy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Parental Communication Intervention | Health Promotion Control Condition. | Total
Number analyzed (Participants) | 330 | 330 | 660
Age, Continuous [Mean (Standard Deviation); unit: Years] — Between 18 and 65 years
  Years
    Adults | 42.41 (8.17) | 42.62 (8.34) | 42.52 (8.25)
    Adolescents | 14.52 (1.26) | 14.57 (1.33) | 14.55 (1.29)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 296 | 295 | 591
  Male | 32 | 35 | 67
  Missing | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 179 | 184 | 363
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 145 | 141 | 286
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 7 | 16
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 42 | 77
  White | 89 | 85 | 174
  More than one race | 24 | 24 | 48
  Unknown or Not Reported | 170 | 170 | 340
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 330 | 330 | 660
Child's Sex [Count of Participants; unit: Participants]
  Female | 174 | 168 | 342
  Male | 154 | 162 | 316
  Missing | 2 | 0 | 2
Marital Status [Count of Participants; unit: Participants]
  Single | 98 | 89 | 187
  Married | 127 | 142 | 269
  Separated | 9 | 13 | 22
  Divorced | 51 | 42 | 93
  Widowed | 5 | 10 | 15
  Live in Partner | 38 | 34 | 72
  Missing | 2 | 0 | 2
Partner [Count of Participants; unit: Participants]
  Yes | 198 | 214 | 412
  No | 129 | 116 | 245
  Missing | 3 | 0 | 3
Education [Count of Participants; unit: Participants]
  Did not complete high school | 32 | 40 | 72
  Completed high school | 95 | 95 | 190
  Did not complete college | 50 | 52 | 102
  Completed college | 151 | 141 | 292
  Missing | 2 | 2 | 4
Employment Outside of Home [Count of Participants; unit: Participants]
  Yes | 128 | 129 | 257
  No | 200 | 201 | 401
  Missing | 2 | 0 | 2
Number of Work Hours per week [Mean (Standard Deviation); unit: Hours] | 33.41 (13.35) | 31.62 (13.35) | 32.50 (13.35)
Average Monthly Income [Count of Participants; unit: Participants]
  <$300 | 22 | 29 | 51
  $300-$799 | 22 | 24 | 46
  $800-$1699 | 24 | 40 | 64
  ≥$1700 | 36 | 18 | 54
  Unknown | 226 | 219 | 445
Government Assistance [Count of Participants; unit: Participants]
  Yes | 210 | 202 | 412
  No | 118 | 128 | 246
  Missing | 2 | 0 | 2
Monthly Government Assistance Income [Mean (Standard Deviation); unit: Currency, US dollars] | 568.78 (854.96) | 537.16 (650.46) | 553.32 (761.09)
Number of Children in House [Mean (Standard Deviation); unit: Child] | 1.53 (0.76) | 1.56 (0.72) | 1.54 (0.74)
Program Location [Count of Participants; unit: Participants]
  Community Agency | 62 | 58 | 120
  School | 172 | 165 | 337
  Home | 46 | 58 | 104
  Other Location | 46 | 46 | 92
  Missing | 4 | 3 | 7
Parents' Computer Comfort [Count of Participants; unit: Participants] — Survey measure to assess parents' comfort with using the computer. Scale used was: very comfortable, somewhat comfortable, somewhat uncomfortable, very uncomfortable.
  Participants
    Very comfortable | 226 | 233 | 459
    Somewhat comfortable | 78 | 73 | 151
    Somewhat uncomfortable | 20 | 15 | 35
    Very uncomfortable | 4 | 7 | 11
    Missing | 2 | 2 | 4
Parents' Ease/Difficulty Finding a Computer [Count of Participants; unit: Participants] — Survey question to measure parents' ease or difficulty in finding a computer to use. Scale was very easy, easy, difficult, very difficult.
  Participants
    Very easy | 140 | 131 | 271
    Easy | 115 | 125 | 240
    Difficult | 52 | 57 | 109
    Very difficult | 20 | 15 | 35
    Missing | 3 | 2 | 5
General Communication between parent and adolescent [Mean (Standard Deviation); unit: Units on a scale] — All items are based on parental self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more communication when talking about general topics. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 3.84 (0.62) | 3.88 (0.59) | 3.86 (0.60)
Sexual Risk Communication between parent and adolescent [Mean (Standard Deviation); unit: Units on a scale] — All items are based on parental self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more communication when talking about sexual risk. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 3.12 (1.12) | 3.31 (1.16) | 3.22 (1.14)
Sexual Prevention Communication between parent and adolescent [Mean (Standard Deviation); unit: Units on a scale] — All items are based on parental self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more communication when talking about sexual prevention. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 3.07 (1.31) | 3.25 (1.35) | 3.16 (1.33)
Sexual Protection Communication between parents and adolescents [Mean (Standard Deviation); unit: Units on a scale] — All items are based on parental self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more communication when talking about sexual protection. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 2.74 (1.36) | 2.93 (1.36) | 2.83 (1.36)
Sexual Peer Pressure between parent and adolescent [Mean (Standard Deviation); unit: Units on a scale] — All items are based on parental self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more communication when talking about sexual peer pressure. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 3.52 (1.21) | 3.71 (1.29) | 3.62 (1.25)
Comfort with Communication between parent and adolescent [Mean (Standard Deviation); unit: Units on a scale] — All items are based on parental self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more comfort with communication. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 3.50 (0.61) | 3.51 (0.60) | 3.5 (0.60)
Sexual Communication Attitudes by adolescents [Mean (Standard Deviation); unit: Units on a scale] — All items are based on adolescent self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more communication when talking about sexual communication attitudes. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 3.71 (0.51) | 3.77 (0.46) | 3.74 (0.49)
Subjective Norms by adolescents [Mean (Standard Deviation); unit: Units on a scale] — All items are based on adolescent self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more communication when talking about subjective norms. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 4.12 (0.79) | 4.19 (0.75) | 4.16 (0.77)
Self-Efficacy by adolescents [Mean (Standard Deviation); unit: Units on a scale] — All items are based on adolescent self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more communication when talking about self-efficacy. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 3.77 (0.90) | 3.89 (0.91) | 3.83 (0.91)
Sexual Communication Intentions by adolescents [Mean (Standard Deviation); unit: Units on a scale] — All items are based on adolescent self-report and measured with 5-point Likert scales (range 1-5), where a higher score indicates more communication when talking about sexual communication intentions. This measure was derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement.
  Units on a scale | 4.02 (0.94) | 4.00 (0.96) | 4.01 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 3 Months in Parent - Adolescent Sexual Risk Communication (Parental Perspective)
Description: Computer-based questionnaire reflecting parent-adolescent sexual risk communication. Data presented from the parental perspective. Questionnaire includes 7 items, each measured using a 5-point Likert scale, ranging from 1-5, where a higher score indicates more communication when talking about sexual topics. All primary outcome measures for this study were derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement. Change was calculated as parent-adolescent sexual risk communication at 3 months minus baseline.
Time Frame: Baseline - 3 months
Population: All participants for whom parent-adolescent sexual risk communication (parental perspective) were recorded at baseline and 3 months.
  Note: for Parental communication intervention arm - 2 missing data points at 3 months); for health promotion arm - 1 missing data at baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parental Communication Intervention | Health Promotion Control Condition.
Number analyzed (Participants) | 255 | 258
units on a scale | 0.54 (.96) | 0.28 (0.81)

2. Primary Outcome: Change From Baseline to 6 Months in Parent - Adolescent Sexual Risk Communication (Parental Perspective)
Description: Computer-based questionnaire reflecting parent-adolescent sexual risk communication. Data presented from the parental perspective. Questionnaire includes 7 items, each measured using a 5-point Likert scale, ranging from 1-5, where a higher score indicates more communication when talking about sexual topics. All primary outcome measures for this study were derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement. Change was calculated as parent-adolescent sexual risk communication at 6 months minus baseline.
Time Frame: Baseline - 6 months
Population: All participants for whom parent-adolescent sexual risk communication (parental perspective) were recorded at baseline and 6 months.
  Note: for health promotion arm - 1 missing data at baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parental Communication Intervention | Health Promotion Control Condition.
Number analyzed (Participants) | 265 | 258
units on a scale | .49 (.95) | .21 (.96)

3. Primary Outcome: Change From Baseline to 12 Months in Parent - Adolescent Sexual Risk Communication (Parental Perspective)
Description: Computer-based questionnaire reflecting parent-adolescent sexual risk communication. Data presented from the parental perspective. Questionnaire includes 7 items, each measured using a 5-point Likert scale, ranging from 1-5, where a higher score indicates more communication when talking about sexual topics. All primary outcome measures for this study were derived as the mean of the individual items, and was calculated for each participant when 75% or more of the items were completed. When less than 75% of the items were completed, the derived measure was considered incomplete and not included in the measurement. Change was calculated as parent-adolescent sexual risk communication at 12 months minus baseline.
Time Frame: Baseline - 12 months
Population: All participants for whom parent-adolescent sexual risk communication (parental perspective) were recorded at baseline and 12 months.
  Note: for health promotion arm - 1 missing data at baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parental Communication Intervention | Health Promotion Control Condition.
Number analyzed (Participants) | 243 | 253
units on a scale | .52 (1.02) | .27 (.97)
Statistical Analysis 1: Comparison: Parental Communication Intervention vs Health Promotion Control Condition; The intervention effect of sexual risk communication (primary outcome in parents) controlling for self-efficacy as a mediator from baseline through 12 months was examined using longitudinal general estimating equations (GEE) modeling, with the Health promotion control condition as the reference category and adjusting for baseline sexual risk communication and average monthly income; Test type: Other — [Not specified]; p = .0229, GEE modeling — Statistical significance taken at the 0.05 level; P-value & estimate rely on group x time interaction effect on primary outcome when controlling for self-efficacy. Used modified Baron & Kenny method; Slope = 0.0153, 95% CI 2-sided [0.0022 to 0.0285], Standard Error of Mean 0.0067 — [Not specified]
Statistical Analysis 2: Comparison: Parental Communication Intervention vs Health Promotion Control Condition; The intervention effect of sexual risk communication (primary outcome in parents) controlling for sexual communication attitudes as a mediator from baseline through 12 months was examined using longitudinal general estimating equations (GEE) modeling, with the Health promotion control condition as the reference category and adjusting for baseline sexual risk communication and average monthly income; Test type: Other — [Not specified]; p = 0.0249, GEE modeling — Statistical significance taken at the 0.05 level; P-value and estimate rely on group x time interaction effect on primary outcome when controlling for sexual communication attitudes. Same method B&K; Slope = 0.0151, 95% CI 2-sided [0.0019 to 0.0282], Standard Error of Mean 0.0067 — [Not specified]
Statistical Analysis 3: Comparison: Parental Communication Intervention vs Health Promotion Control Condition; The intervention effect of sexual risk communication (primary outcome in parents) controlling for subjective norms as a mediator from baseline through 12 months was examined using longitudinal general estimating equations (GEE) modeling, with the Health promotion control condition as the reference category and adjusting for baseline sexual risk communication and average monthly income; Test type: Other — [Not specified]; p = 0.0204, GEE modeling — Statistical significance taken at the 0.05 level; Reported P-value and estimate rely on the group x time interaction effect on primary outcome when controlling for subjective norms. Same method B&K; Slope = 0.0158, 95% CI 2-sided [0.0025 to 0.0292], Standard Error of Mean 0.0068 — [Not specified]

ADVERSE EVENTS:
Arm/Group | Parental Communication Intervention | Health Promotion Control Condition.
Serious Adverse Events (participants affected / at risk) | 0/330 | 0/330
Other Adverse Events (participants affected / at risk) | 0/330 | 0/330

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-06-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT03063385/Prot_000.pdf